CLINICAL TRIAL: NCT05111197
Title: Local Ablative Stereotactic Radiotherapy for Residual Hypermetabolic Lesion in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer Long-term Responders to Immunotherapy : a Randomized, Multicenter, Open-label Phase III Study
Brief Title: Local Ablative Stereotactic Radiotherapy for Residual Hypermetabolic Lesion in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer Long-term Responders to Immunotherapy
Acronym: TRAILOCLORI01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2021-08
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-02

CONDITIONS: Locally Advanced Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer
Keywords: lung; Immunotherapy; Stereotactic radiotherapy; 18F- FDG PET/ CT; Locally advanced cancer; Metastatic cancer; Overall survival; Progression Free Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A. (Immunotherapy + SRT) (Experimental): Continuation of anti-PD-1 or anti-PD-L1 immunotherapy, started at least 6 months ago, associated with Stereotactic Radiation Therapy (SRT)
  Interventions: Radiation: SRT; Drug: Immunotherapy
- B (Immunotherapy alone) (Active Comparator): Continuation of anti-PD-1 or anti-PD-L1 immunotherapy alone (started at least 6 months ago)
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Radiation: SRT — Patients with a maximum of 5 residual hypermetabolic lesions observed on 18F- FDG PET / CT after a minimum of 6 months of immunotherapy are treated with SRT, in addition to their anti-PD-1 or anti-PD-L1 immunotherapy as it was administered before randomization in the trial, according to the standards.
  A maximum of 3 Brain metastases treatable in stereotactic radiotherapy will be included among these hypermetabolic lesions.
  Each lesion is treated with a total dose of 24 Gy delivered in 3 fractions of 8 Gy (isodose surface).
  Arms: A. (Immunotherapy + SRT)
Drug: Immunotherapy — Patients with a maximum of 5 residual hypermetabolic lesions observed on 18F- FDG PET / CT after a minimum of 6 months of immunotherapy continue their anti-PD-1 or anti-PD-L1 immunotherapy as it was administered before randomization in the trial, according to the standards.

SUMMARY:
At present, it is recommended to continue immunotherapy until progression or unacceptable toxicity.

However, only a minority of patients benefits from a durable response and most see the disease progress despite several months of control under immunotherapy. Multimodal approaches have been developed to improve their prognosis.

This study, randomized, open-label study aims to evaluate the impact of addition of ablative radiotherapy on OS of patients with NSCLC and oligometastatic lesions and treated by immunotherapy in first line (potentially associated with chemotherapy) or beyond. Stereotactic radiotherapy will be performed on a maximum of 5 residual hypermetabolic lesions seen on 18F-FDG PET / CT, in patients responding to immunotherapy (or with a stable disease) for at least 6 months.

DETAILED DESCRIPTION:
Description of the modalities for recruiting :

During a standard consultation, the oncologist presents the study to the patient with locally advanced or metastatic non-small cell lung cancer long-term responders to immunotherapy. He gives the patient the consent form to participate in the study.

Once the consent form has been signed by the patient and the investigator, the investigator prescribes a screening test which must be carried out within 30 days before the randomization (Day 0, D0).

The screening step includes in particular a complete physical exam, a clinical laboratory tests a thoraco abdomino pelvic (TAP) and cerebral CT scan, a cerebral MRI (for patients with cerebral lesions observed on cerebral CT scan), a Spinal MRI (for patients with bones lesions observed on TAP CT scan), a PET scan (18F-FDG) (the results will be routinely interpreted in the centre and will be centrally reviewed), Patient Reported Outcome (PRO), QLQ-C30 and QLQ LC13

The inclusion of a patient is conditioned by the following definitive criterion : Maximum 5 residual hypermetabolic lesions measured on the CT from the 18F-FDG PET / CT centrally reviewed, including primary tumor and a maximum of 3 brain asymptomatic metastases (even if they are poorly seen in 18F- FDG PET/CT) treatable in stereotactic radiotherapy.

Patients registration and randomization :

Any patient who has signed an informed consent form (ICF) must be registered in the eCRF in order to be assigned a patient number.

Randomization will be centralized and performed via the eCRF. Patients will be randomly assigned (1:1) to either continuation of immunotherapy alone or addition of local ablative radiotherapy to immunotherapy.

The randomization procedure using minimization method will be stratified by the investigation center, by the treatment line (1 vs ≥2) and by the immunotherapy (pembrolizumab and nivolumab versus atezolizumab).

Treatment period :

Both arms continue the anti-PD1 or anti-PDL-1 immunotherapy according to the medical prescription.

Arm A (experimental), SRT start maximum 3 weeks after randomisation

Follow-up visits include in particular a complete physical exam, a clinical laboratory tests, a thoraco abdomino pelvic and cerebral CT scan, a cerebral MRI (for patients with cerebral lesions observed on cerebral CT scan), a Spinal MRI (for patients with bones lesions observed on TAP CT scan), a PET scan (18F-FDG) at 6 months post-randomization only (the results will be routinely interpreted in the centre and will be centrally reviewed) ; Patient Reported Outcome (PRO), QLQ-C30 and QLQ LC13

Imaging surveillance (CT scan +/- cerebral MRI +/- spinal MRI) will be performed for each patient up to progression or up to 12 months after randomization of the last patient included in the absence of progression.

Vital status is collected once a year and also date of death if applicable for each patient up to 12 months after randomization of the last patient included.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or more,
* Patient treated for histologically proven non-small cell lung cancer,
* Stage IIIB or IV,
* Performance status 0 to 2,
* Patient treated by immunotherapy (anti PD-1 or anti PD-L1) started for at least 6 months and regardless of the treatment line (in first line, immunotherapy may have been combined with chemotherapy),
* Response or stable disease on thoraco abdomino pelvic and cerebral CT scan,
* Maximum 5 residual hypermetabolic lesions measured on the 18F-FDG PET / CT centrally reviewed, including primary tumor and a maximum of 3 asymptomatic brain metastases (even if they are poorly seen in 18F- FDG PET/CT) treatable in stereotactic radiotherapy (extracerebral lesions ≤ 4cm and brain lesions ≤ 3cm measured on CT scanners)
* Effective contraception used in women of childbearing potential
* Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations,
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up,
* Patient has valid health insurance.

Exclusion Criteria:

* Persistence of grade 2 or greater adverse effects of immunotherapy,
* Infection in progress,
* At least one of the 5 hypermetabolic lesions measured on the 18F-FDG PET / CT centrally reviewed in a previously irradiated area,
* Uncontrolled severe comorbidity,
* History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥ 3 years and of low potential risk for recurrence ; Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease ; Adequately treated carcinoma in situ without evidence of disease
* Pregnant or nursing patient
* Patient deprived of liberty or under guardianship,
* Patient unable to undergo regular medical check-ups for geographical, social or psychological reasons.
* Disorder precluding understanding of trial information or informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The overall survival (OS) benefit of local treatment by stereotactic radiotherapy with immunotherapy versus immunotherapy alone | 12 months post-randomization
  Overall survival rate, where OS is the time between randomization and death of any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 12 months after randomization of the last patient included
  Median overall survival at the end of the study
Progression Free Survival (PFS) | 12 months after randomization of the last patient included
  Median PFS, time between randomization and progression or death in absence of progression, at the end of the study
Quality of life (Qol) | 12 months after randomization
  EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30)
Quality of life (Qol) | 12 months after randomization
  Lung cancer-specific Quality of Life Questionnaire EORTC QLQ-LC13
Overall survival (OS) in patients with complete metabolic response rate on 18F- FDG PET / CT 6 months after randomization | 6 months after randomization in the SRT arm
  Median overall survival at the end of the study in patients with complete metabolic response rate on 18F- FDG PET / CT (PERSIST)
Progression Free Survival (PFS) according to complete metabolic response rate on 18F- FDG PET / CT 6 months after randomization | 6 months after randomization in the SRT arm
  Median PFS at the end of the study in patients with complete metabolic response rate on 18F- FDG PET / CT (PERSIST) 6 months after randomization in the SRT arm

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - ICO - Site Paul Papin, Angers
  - Chu de Brest, Brest
  - Centre François BACLESSE, Caen
  - Institut de cancérologie de l'ouest, Saint-Herblain
  - Chu de Tours, Tours